CLINICAL TRIAL: NCT06099899
Title: Qualitative Study on Factors Impeding Physical Activity During the Post-discharge Period After Hematopoietic Stem Cell Transplantation in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-972-01
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Physical Activities
Keywords: hematopoietic stem cell transplantation
MeSH Terms: conditions — Motor Activity | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- child: The child's age ranges from 8 to 18 years old. They have undergone hematopoietic stem cell transplantation for at least one month. They do not have any mental disorders or consciousness impairments. The child is capable of independent walking. The interviewees are able to express their thoughts clearly.
  Interventions: Other: interview
- parent: The primary caregivers during the home care period for these children.
  Interventions: Other: interview

INTERVENTIONS:
Other: interview — conduct in-depth interviews

SUMMARY:
The purpose is to gain a deep understanding of the hindering factors in physical activities during the home period after pediatric hematopoietic stem cell transplantation, in order to provide references for developing targeted intervention measures.

DETAILED DESCRIPTION:
From October 2023 to September 2024, a purposive sampling method will be used to select 10 post-pediatric hematopoietic stem cell transplant patients and 10 family members receiving treatment at Sun Yat-sen Memorial Hospital, Zhongshan University, as the subjects for the study. The phenomenological approach in qualitative research will be employed to conduct in-depth interviews with them, and data analysis will be performed using the Colaizzi analysis method.

ELIGIBILITY:
Inclusion Criteria:

* The child's age ranges from 8 to 18 years old.
* They have undergone hematopoietic stem cell transplantation for at least one month.
* They do not have any mental disorders or consciousness impairments.
* The child is capable of independent walking.
* The interviewees are able to express their thoughts clearly.
* Both the child and their family members are informed about and have given consent to participate in this study.

Exclusion Criteria:

* Relapse or the presence of other tumors
* Physical activity prohibitions, such as movement disorders, platelet count <20×10⁹, -acute bleeding, hemoglobin level <80g/L
* Fever with a temperature of 38.8℃ or higher due to infection
* Pain score of 4 or higher
* Other severe complications, such as heart failure or severe malnutrition.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children during the post-hematopoietic stem cell transplantation period at home
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the hindering factors in physical activities interview | 2 month
  Colaizzi analysis method

CONTACTS AND LOCATIONS:
Overall Officials: QIAN HAO, nurse, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No